CLINICAL TRIAL: NCT05181462
Title: A Randomized Non-comparative Open-label Phase 1b/2 Study of Nadunolimab in Combination with Gemcitabine Plus Carboplatin in Patients with Advanced Triple Negative Breast Cancer. "TRIFOUR Study"
Brief Title: Nadunolimab in Combination with Gemcitabine Plus Carboplatin in Patients with Advanced Triple Negative Breast Cancer.
Acronym: TRIFOUR
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cantargia AB (Industry)
Collaborators: Spanish Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAN04CLIN005; 2021-003402-46 (EudraCT Number)
Record Dates: First submitted 2021-12-01; First posted 2022-01-06 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Triple Negative Breast Cancer
Keywords: Unresectable locally advanced; Metastatic triple negative breast cancer; Nadunolimab
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Carboplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Phase Ib: Single-arm (dose-escalation 3+3 design).
  * Nadunolimab escalation (Dose Level (DL) -1: 0.5 mg/Kg, DL 1: 1 mg/kg, DL 2: 2.5 mg/kg), DL 3: 5 mg/kg IV on days 1 and 8/15, in cycles of 3-4 weeks.
  * Gemcitabine 1000 mg/m2 IV on days 1 and 8/15, in cycles of 3-4 weeks.
  * Carboplatin Area Under the Curve (AUC) 2 mg/mL/min intravenous (IV) on days 1 and 8/15, in cycles of 3-4 weeks.
  Phase II: Randomized 1:1, non-comparative, open-label.
  Patients randomized to arm A will receive:
  * Nadunolimab Recommended Phase II Dose (RP2D) mg/kg IV on days 1 and 8/15, in cycles of 3-4 weeks.
  * Gemcitabine 1000 mg/m2 IV on days 1 and 8/15, in cycles of 3-4 weeks.
  * Carboplatin AUC 2 mg/mL/min IV on days 1 and 8/15, in cycles of 3-4 weeks.
  Patients randomized to arm B will receive:
  * Gemcitabine 1000 mg/m2 IV on days 1 and 8/15, in cycles of 3-4 weeks.
  * Carboplatin AUC 2 mg/mL/min IV on days 1 and 8/15, in cycles of 3-4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase Ib: Single-arm (dose-escalation 3+3 design). (Experimental): * Carboplatin Area Under the Curve (AUC) 2 mg/mL/min intravenous (IV) on days 1 and 8, every 3-week cycles.
  * Gemcitabine 1000 mg/m2 IV on days 1 and 8, every 3-week cycles.
  * Nadunolimab escalation (DL -1: 0.5 mg/Kg, DL 1: 1 mg/kg, DL 2: 2.5 mg/kg), DL 3: 5 mg/kg IV on days 1 and 8, every 3-week cycles.
  Interventions: Drug: Carboplatin; Drug: Gemcitabine; Drug: Nadunolimab
- Phase II: Randomized 1:1, non-comparative, open-label.Patients randomized to arm A (Experimental): * Carboplatin AUC 2 mg/mL/min IV on days 1 and 8, every 3-week cycles.
  * Gemcitabine 1000 mg/m2 IV on days 1 and 8, every 3-week cycles.
  * Nadunolimab Recommended Phase II Dose (RP2D) mg/kg IV on days 1 and 8, every 3-week cycles
  Interventions: Drug: Carboplatin; Drug: Gemcitabine; Drug: Nadunolimab
- Phase II: Randomized 1:1, non-comparative, open-label.Patients randomized to arm B (Active Comparator): * Carboplatin AUC 2 mg/mL/min IV on days 1 and 8, every 3-week cycles.
  * Gemcitabine 1000 mg/m2 IV on days 1 and 8, every 3-week cycles.
  Interventions: Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Carboplatin — Carboplatin Area Under the Curve (AUC) 2 mg/mL/min intravenous (IV) on days 1 and 8/15, in cycles of 3-4 weeks
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 IV on days 1 and 8/15, in cycles of 3-4 weeks
Drug: Nadunolimab — Nadunolimab escalation (DL -1: 0.5 mg/Kg, DL 1: 1 mg/kg, DL 2: 2.5 mg/kg), DL 3: 5 mg/kg IV on days 1 and 8/15, in cycles of 3-4 weeks.
  Other Names: CAN04
  Arms: Phase II: Randomized 1:1, non-comparative, open-label.Patients randomized to arm A; Phase Ib: Single-arm (dose-escalation 3+3 design).

SUMMARY:
Triple negative breast cancer (TNBC) represents approximately 15% of all breast cancers (BC) worldwide. The term triple negative means that tumor growth is not stimulated by the hormones estrogen and progesterone, nor by the HER2 protein, so unlike other types of BC, TNBC, which is an aggressive form of BC, does not have specific effective therapies available being the least common form of BC and the most difficult to treat.

Advanced or metastatic TNBC is treated with combinations of platinum-based chemotherapy with taxanes or gemcitabine with a 5-year survival rate of 12%. Recent studies have shown that TNBC expresses Interleukin 1 Receptor Accessory Protein (IL1RAP) at higher levels than other forms of BC.

Nadunolimab is a fully humanized monoclonal antibody that blocks the signals that occur within the cell produced by IL1RAP protein, thereby impairing the cancer cells' ability to secrete tumor stimulating substances, in turn reducing the tumor, inflammation and tumor progression. On the other hand, it is an antibody designed to activate the immune system to fight cancer cells.

This clinical trial is divided into two phases, phase Ib in which it is expected to include up to 15 patients and phase II in which it is expected to include 102 patients. The main purpose of phase Ib is to ensure that the combination of nadunolimab plus chemotherapy (gemcitabine plus carboplatin) is safe and determine the highest dose of nadunolimab that can be given safely without causing serious side effects. If the pre-specified objectives in this part are achieved, the trial will be expanded to a randomized phase II, to evaluate the efficacy of the combination of nadunolimab plus gemcitabine plus carboplatin, compared to a control group that will receive gemcitabine plus carboplatin only.

DETAILED DESCRIPTION:
Triple negative breast cancer (TNBC) represents approximately 15% of all breast cancers worldwide and is characterized by the absence of estrogen receptor (ER), progesterone receptor (PR), and human epidermal growth factor receptor 2 (HER2) expression. TNBC is more common in African American women, in premenopausal women and in BRCA1/2 mutation carriers. TNBC presents the worst outcomes of all breast cancer (BC) subtypes with a 5-year overall survival (OS) of 78.5%, even when the analyses are adjusted for age, disease stage, race, tumor grade and adjuvant chemotherapy (CT). One in three TNBC patients will develop distant metastases, which typically occurs within the first 3 years of initial diagnosis, and persistently, one in five TNBC patients will succumb to their metastatic disease in less than 5 years. The 5-year survival rates for localized, regional, and metastatic TNBC are 91%, 65%, and 12% , respectively. The dismal prognosis of high-risk, locally advanced and metastatic TNBC highlights an unmet need for an improved survival in these patients. Another reason for the poor outcomes associated with TNBC is the lack of effective targeted therapies. As a result, standard cytotoxic CT remains the backbone of systemic therapy in TNBC patients.

Further attempts to classify TNBC into distinct subtypes based on unique tumor/tumor microenvironment (TME) cellular signatures and messenger ribonucleic acid (mRNA) expression profiles may provide relevant information about the molecular drivers, actionable therapeutic targets and effective therapy selection. Based on the PAM50 gene expression profile, 78.6% of TNBC have significant overlap with the basal-like molecular subtype. The remaining gene expression profiles of TNBC (21.4%) may be further subclassified as normal-like (7%), HER2-enriched (7.8%), luminal B (4.4%), and luminal A (2.2%). Even though the assessment and characterization of TNBC into molecular subtypes is not currently performed clinically on a routine basis, these sub-classifications based on unique cellular signatures and global RNA expression profiles may provide therapeutic insights for each specific subset of TNBC patients.

Current available treatments for advanced TNBC are palliative in nature and are based mostly on the use of cytotoxics. Recently poly Adenosine diphosphate (ADP) ribose polymerase inhibitors (PARPi), (olaparib, talazoparib) have shown efficacy in patients with germline BRCA (gBRCA) mutant tumors, with olaparib and talazoparib already approved in the advanced setting. Atezolizumab in combination with nab-paclitaxel has been approved for patients with unresectable locally advanced or metastatic TNBC whose tumors express programmed death-ligand 1 (PD-L1). Pembrolizumab, in combination with CT (paclitaxel, or nab-paclitaxel, or gemcitabine plus carboplatin), has been granted accelerated approval by the Food and Drug Administration (FDA) for locally recurrent unresectable or metastatic TNBC not previously treated with CT in the metastatic setting and with PD-L1 expression (Combined Positive Score (CPS) ≥ 10) as determined by the PD-L1 immunohistochemistry (IHC) 22C3 pharmDx (Dako North America, Inc.), also approved by the FDA as a companion diagnostic. Despite of these interesting results, new treatments are necessary for patients with TNBC.

Platinum agents have recently become an important treatment option in the management of TNBC, especially in patients with BRCA mutations or PD-L1-negative or who have progressed to immune checkpoint inhibitors, as carboplatin demonstrated comparable efficacy and a more favorable toxicity profile compared with docetaxel. Platinum-based regimens are particularly appealing in TNBC based on their DNA-damaging mechanism of action , due to the high genomic instability observed on this type of BC, particularly in patients harbouring gBRCA1/2 mutations or "BRCAness" (homologous recombination repair defects in the absence of gBRCA1/2 mutations). The TNT trial showed that carboplatin is a particularly active drug in gBRCA mutated BC patients. In the metastatic setting, interesting activity has been reported with the gemcitabine plus carboplatin combination (dose of 1,000 mg/m2 and area under the curve [AUC] 2 mg x min/mL, respectively, on days 1 and 8 of each 3-week cycle), in both phase II and III trials testing the role of iniparib in advanced TNBC with a median progression-free survival (PFS) of 3.1 and 4.1 months, and a median OS of 7.7 and 11.1 months, respectively. In exploratory analyses by line of therapy in the phase III trial, patients who received first line treatment had a median PFS of 4.6 months and a median OS of 12.6 months; for those patients treated in second line, the median PFS was 2.9 months and the median OS was 8.1 months. Regarding the tumor response according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 with confirmation of response and independent central review, the following percentages were reported: a) complete response (CR) 1.6%; b) partial response (PR) 29%; c) stable disease (SD) 35% (lasting more than 6 months in 5.4%); d) progressive disease (PD) 24%; and e) nonevaluable 5.4%. The overall response rate (ORR) was 30% (95% Confidence Interval (CI), 25-36%) and the clinical benefit rate (CBR) with SD > 6 months, 36%. If we consider the Treatment Emergent Adverse Events (TEAEs) published in 2014, the most frequent AEs included neutropenia 65% (Grade [G] 3/4 53%), fatigue 63% (G 3/4 6%), anemia 62% (G 3/4 22%), nausea 59% (G 3/4 3%), thrombocytopenia 54% (G 3/4 24%), constipation 42% (G 3/4 < 1%), and vomiting 31% (G 3/4 1%). Data from the tnAcity trial in the first line setting showed a median PFS of 6.0 months and a median OS of 12.6 months in the control arm treated with gemcitabine 1,000 mg/m2 plus carboplatin AUC 2 mg x min/mL, on days 1 and 8 of 3-week cycles. Another efficacy results published include the 12-month PFS rate (11%), ORR (44% [CR 8%, PR 36%]), median duration of response (DoR) (5.0 months), SD ≥ 4 months (32%), PD as best response (21%). At least one G ≥ 3 AE was reported in 84% of patients and at least one serious AE in 39% of patients with this combination. The most frequently observed G ≥ 3 AEs were neutropenia (52%), thrombocytopenia (28%), anemia (27%), leukopenia (11%), fatigue (3%) and peripheral neuropathy (2%). The meta-analysis with data from more than 4,500 patients supports the use of platinums in Advanced Breast Cancer (ABC) and this recommendation is considered in current international practice guidelines ABC.

ELIGIBILITY:
Inclusion Criteria: Patients are eligible to be enrolled in the study only if they meet all of the following criteria:

1. The patient has signed and dated the informed consent form (ICF) and it has been obtained before conducting any specific procedure for the study.
2. Female or male BC patients of ≥ 18 years of age.
3. Permission to access archived tumor tissue sample (either from primary breast tumor or a metastatic lesion, preferably the most recent one) for biomarker analysis. Not having archived tissue is not a reason to exclude the patient from enrollment.
4. Paired tumor biopsies, pre-treatment and on-treatment, for pharmacodynamic analysis are not compulsory and will be obtained as per investigator judgement and patient decision. However, patients and investigators are encouraged to obtain them if the patient has easily accessible disease like skin or superficial lymph nodes. Ideally, the same lesion (always in the same organ) should be biopsied before treatment and on treatment whenever possible. It is allowed to use archived biopsies as pre-treatment samples, obtained after ending the previous systemic treatment).
5. The lesion accessible for biopsy may not be the only target lesion and should not be located in a previously irradiated field (unless this index lesion has PD ≥ 20% post-radiation).
6. Histologically confirmed TNBC that is either locally recurrent, inoperable and cannot be treated with curative intent or is metastatic:

   1. Documented Hormone Receptor (HR) negative BC based on local laboratory determination on the most recent tumor biopsy. HR negative defined as < 1% positive cells by immunohistochemistry (IHC) for estrogen receptor (ER) and progesterone receptor (PgR).
   2. Documented Human Epidermal Growth Factor Receptor 2 (HER2) negative BC based on local laboratory determination on the most recent tumor biopsy. HER2 negative tumor is determined according to recommendations of the applicable American Society of Clinical Oncology (ASCO)/ College of American Pathologists (CAP) guidelines available.
   3. Patients are eligible for the study irrespectively of BRCA1/2 mutational status. It is not required to have the analysis performed before the study inclusion.
7. Patients should be eligible to receive gemcitabine and carboplatin as the following line of therapy. No more than 1 previous line of systemic therapy for the advanced disease is allowed:

   1. Those patients with PD during or within 6 months after completing the (neo)adjuvant treatment are allowed to be included in the study and are considered for second-line group of patients.
   2. Prior therapy with immuno-checkpoint inhibitors (ICIs) either in the metastatic setting (as first-line therapy) or in the (neo)adjuvant setting is allowed.
   3. Previous treatment with platinum-derived agents in early-stage setting is allowed if the platinum-free interval is at least of 12 months.
   4. Prior therapy with PARP inhibitors is allowed.
8. Documented progressive disease (i.e. biopsy sample, pathology or imaging report) from the last treatment.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
10. Patients must have at least one measurable lesion that can be accurately assessed at baseline and is suitable for repeated assessment by CT scan, MRI, plan X-ray or physical examination. Clinical lesions will only be considered measurable when they are superficial and ≥ 10mm in diameter as assessed using callipers (e.g. skin nodules). Patients with bone-only disease must have a lytic or mixed (lytic + blastic) lesion, which has not been previously irradiated and can be accurately assessed by CT scan/MRI according to RECIST version 1.1 (with a component of soft tissue mass).
11. Adequate organ and bone marrow function defined as follows:

    1. Absolute Neutrophil Count (ANC) ≥ 1.500/mm3 (1.5x109/L), without previous Granulocyte Colony-Stimulating Factor (G-CSF) within 2 weeks prior to the study treatment.
    2. Platelets ≥ 100.000/mm3 (100x109/L), without previous transfusion within 2 weeks prior to the study treatment.
    3. Hemoglobin ≥ 9 g/dL (90 g/L), without previous transfusion within 28 days before starting with the study treatment.
    4. Serum creatinine ≤ 1.5 x Upper Limit of Normal (ULN) or estimated creatinine clearance ≥ 60 mL/min as calculated using the Cockcroft-Gault formula.
    5. Total serum bilirubin ≤ 1.5 x ULN (≤ 3.0 x ULN if Gilbert´s disease).
    6. Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT) ≤ 3.0 x ULN (≤ 5.0 x ULN if liver metastases present).
    7. Alkaline phosphatase ≤ 2.5 x ULN (≤ 5.0 x ULN if bone or liver metastases present).
12. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE v5.0 Grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion). In case of immune-related toxicities, adequately resolved to Grade 1 or non-persistent Grade 2 AEs with the recommended measures by the current guidelines.
13. Patients testing positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must meet ALL the following criteria:

    1. Have CD4+ T-cell (CD4+) counts ≥ 350 cells/µL.
    2. Have not had an opportunistic infection within the past 12 months. Patients on prophylactic antimicrobials can be included in the study.
    3. Should be on stable antiretroviral therapy for at least 4 weeks.
    4. Have an HIV viral load less than 400 copies/mL prior to enrolment.
14. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
15. Negative serum pregnancy test within 7 days prior to enrolment for premenopausal women, and for women who have experienced menopause onset < 12 month prior to first dose of therapy..

    * For premenopausal women: agreement to remain abstinent or use single or combined non-hormonal contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 7 months after the last dose of study treatment.
    * For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and to refrain from donating sperm during the same period, as defined below with female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose of carboplatin/gemcitabine to avoid exposing the embryo. Due to the possibility of irreversible infertility with carboplatin/gemcitabine, men receiving these chemotherapies should consult with their doctor regarding conservation of sperm prior to treatment initiation.

Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Examples of non-hormonal contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide.

Exclusion Criteria:Patients will be excluded from the study if they meet any of the following criteria:

1. Patient has received extended field radiotherapy ≤ 4 weeks before the start of treatment (≤ 2 weeks for limited field radiation for palliation), and who has not recovered to ≤ Grade 1, according to NCI CTCAE v5.0, from related AEs of such therapy (except for alopecia).
2. Treatment with systemic anticancer treatments, investigational products, or major surgery within 4 weeks before the first dose of study drug or 5 half-lives, whichever is shorter. Patients should have recovered from previous treatment toxicity to ≤ Grade 1 (except alopecia and peripheral neuropathy).
3. No prior treatment with an anthracycline and a taxane unless contraindicated or not considered the most suitable treatment option (e.g. in the de novo metastatic setting) according to physician's opinion.
4. Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction, or cerebrovascular accident within 3 months prior to randomization, unstable arrhythmias, or unstable angina. Patients with a known left ventricular ejection fraction (LVEF) < 50% will be excluded.
5. Patients with known coronary artery disease or congestive heart failure (CHF) not meeting the above criteria, must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
6. Presence of an abnormal ECG that is clinically significant in the investigator's opinion, including complete left bundle branch block, second or third-degree heart block, or QT interval corrected using Fridericia's formula (QTcF) > 480 ms demonstrated by at least two consecutive ECGs.
7. Patients with uncontrolled brain metastases; however, patients who have been previously treated with surgery, whole-brain radiation, and/or stereotactic radiosurgery and are considered controlled (with ≤ 10 mg/day of prednisone or equivalent) at the time of receiving the first dose of nadunolimab are allowed. For asymptomatic patients, screening brain imaging is not required.
8. Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to enrolment.
9. Severe (Grade 3) infection requiring oral or IV antibiotics within 4 weeks prior to enrolment, including but not limited to hospitalization for complications of infection, bacteremia, or pneumonia. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
10. Positive hepatitis B surface antigen (HBsAg) test at screening: Total hepatitis B core antibody (HBcAb) test at screning must be negative. If HBsAg and HBcAb are positive, hepatitis B virus (HBV) DNA test at screening should be performed and if patient does not have viral load, patient can be enrolled into the study.
11. Positive hepatitis C virus (HCV) antibody test at screening: if positive, HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
12. Pregnant or lactating or intending to become pregnant during or within 6 months after the last dose of study treatment.
13. Known hypersensitivity or allergy to any component of the nadunolimab, carboplatin or gemcitabine drug formulations, and known hypersensitivity to platinum-containing compounds.
14. Patients who receive a live vaccination, etanercept, or other Tumor necrosis factor (TNF)-alpha inhibitors just prior to participation in this study (within 28 days of first study drug administration).
15. Patients with a history of autoimmune disease requiring systemic immunosuppressive therapy (daily prednisone equivalent doses > 10 mg/day). Patients with autoimmune diseases and without systemic therapies are allowed.
16. Diagnosis of any other malignancy within 5 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of any origin or stage I colorectal.
17. Patients with a history of slowly progressive dyspnea and non-productive cough or disorders such as sarcoidosis, silicosis, idiopathic pulmonary fibrosis, hypersensitivity pneumonitis lung or multiple allergies.
18. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
19. Polymerase chain reaction (PCR) positive or antigen test positive for coronavirus disease 2019 (COVID-19). Patients who had previously symptomatic COVID-19 infection should have recovered to Grade ≤ 1 or baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of Dose Limiting Toxicity (DLT) within the first cycle of nadunolimab in combination with gemcitabine plus carboplatin | At the end of Cycle 1 (each cycle is 21 days)
  DLT is defined according to the NCI-CTCAE version 5.0 as any of the following events considered by investigator to be related to investigational treatment:
  1. Grade (G) 5 Treatment Emergent AE
  2. G ≥ 3 neutropenia + fever and/or infection (single temp. > 38.3°C or sustained temp. ≥ 38°C >1 hour)
  3. G 4 neutropenia > 7 days
  4. G 4 thrombocytopenia > 3 days
  5. G ≥ 3 thrombocytopenia > 7 days or accompanied by G 2 bleeding or platelet transfusion
  6. Delay in the initiation of Cycle 2 > 14 days from the calculated start date due to a lack of adequate recovery of treatment-related hematological or non-hematological toxicity
  7. G ≥ 3 AE with permanent discontinuation of any of the study drugs
  8. Elevations of bilirubin and transaminases meeting Hy's Law criteria
  9. G 4 laboratory abnormalities discussed with the Medical Coordinators, Sponsor and GEICAM
  10. G ≥ 3 non-hematological toxicity
  11. G 2 toxicity considered a dose limiting
Objective Response Rate (ORR) | Through study completion, an average of 58 months
  Tumor response is assessed according to Response Evaluation Criteria for Solid Tumors (RECIST) version 1.1 as per investigators' assessment.
  ORR is defined as the rate of Complete Response (CR) plus Partial Response (PR) according to RECIST version 1.1, out of the patients who receive at least one dose of treatment and have measurable disease. These results will be calibrated against the ORR in the control arm.

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | Through study completion, an average of 58 months
  CBR is defined as the rate of a Complete Response (CR) plus Partial Response (PR) plus Stable Disease (SD) lasting ≥ 24 weeks, according to RECIST v1.1 and as per investigator's assessment out of enrolled patients. n. Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions; SD is defined as a failure to meet criteria for CR or PR in the absence of progressive disease
Disease Control Rate (DCR) | Through study completion, an average of 58 months
  DCR is defined as the rate of CR, PR plus SD of any duration, according to RECIST v1.1 and as per investigator's assessment out of enrolled patients.
Duration of Response (DoR) | Through study completion, an average of 58 months
  DoR assessed according to RECIST v1.1, is defined as the time from the date of first documentation of overall response (CR or PR) to the date of first documented progressive disease (PD), or death from any cause, whichever occurs first. PD is defined using RECIST, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Progression-Free Survival (PFS) | Through study completion, an average of 58 months
  PFS according to RECIST v1.1 as per the investigator's assessment. It is defined as the time from the date of enrolment to the date of PD or death from any cause, whichever occurs first.
Proportion of patients free of PD at 6 and 12 months | Up to 12 months
  PD is defined using RECIST, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions within 6 and 12 months.
PFS rate at 6 and 12 months | Up to 12 months
  PFS according to RECIST v1.1 as per the investigator's assessment. It is defined as the time from the date of enrolment to the date of PD or death from any cause, whichever occurs first at 6 and 12 months
Overall Survival (OS) | Through study completion, an average of 58 months
  OS is defined as the time from the date of enrolment to the date of death from any cause.
Proportion of patients alive at 12 and 18 months | Up to 12 months
  Proportion of patients alive at 12 and 18 months; based on the median duration of OS observed.
Immune Overall Response Rate (iORR) | Through study completion, an average of 58 months
  Response parameters per Guidelines for Response Criteria for Use in Trials Testing Immunotherapeutics (iRECIST) criteria in patients who receive treatment beyond PD by RECIST 1.1 Tumor response is assessed using iRECIST. iORR is defined as the percentage of patients with a Immune Complete Response (iCR) or Immune Partial Response (iPR) out of the patients from the efficacy population. Per iRECIST, iCR is defined as the disappearance of all measurable and non-measurable lesions, and lymph nodes must decrease to < 10 mm in short axis; iPR is defined as an >=30% decrease in total measured tumor burden relative to baseline; Immune Overall Response (iOR) = iCR + iPR.
Immune Clinical Benefit Rate (iCBR) | Through study completion, an average of 58 months
  Response parameters per iRECIST criteria in patients who receive treatment beyond PD by RECIST 1.1 Tumor response is assessed using iRECIST. iCBR is defined as the rate of a Immune Complete Response (iCR) plus Immune Partial Response (iPR) plus Immune Stable Disease (iSD) lasting ≥ 24 weeks iCR is defined as the disappearance of all target lesions; iPR is defined as an >=30% decrease in the sum of the longest diameter of target lesions; iSD is defined as a failure to meet criteria for iCR or iPR in the absence of progressive disease
Immune Disease Control Rate (iDCR) | Through study completion, an average of 58 months
  Response parameters per iRECIST criteria in patients who receive treatment beyond PD by RECIST 1.1 iDCR is defined as the rate of iCR, iPR plus iSD of any duration
Immune Progression Free Survival (iPFS) | Through study completion, an average of 58 months
  Response parameters per iRECIST criteria in patients who receive treatment beyond PD by RECIST 1.1 iPFS is defined as the time from the date of enrolment to the date of immuno Progressive Disease (iPD) or death from any cause, whichever occurs first.
The Number of Participants Who Experienced Adverse Events (AE) | Through study completion, an average of 58 months
  It will be assessed by the frequency, severity and nature of AEs, serious adverse event (SAE), changes in vital signs and standard clinical and laboratory tests (haematology, serum chemistry, and urine). The severity of AEs will be graded by the NCI CTCAE version 5.0 and the AE terms will be coded by the current version of the Medical Dictionary for Regulatory Activities (MedDRA).
Change from baseline (CFB) by Quality of Life (QoL) | At 12,18 and 24 months
  CFB in the global health status (GHS) score and each scale of the EORTC quality of life questionnaire (QLQ) -C30 questionnaire.
  Patient reported outcomes of health-related quality of life will be assessed using the EORTC QLQ-C30 questionnaire and analyzed on the QoL population.
  Published scoring manuals and guidelines will be used to generate scale scores and handle missing data. Descriptive statistics for actual values will be tabulated at each scheduled time point.
  CFB will be presented at each scheduled time point for the GHS score and each of the functionals and symptoms scales from the EORTC QLQ-C30 questionnaires.
  Longitudinal analysis of scores will be performed using linear mixed models.
Time to deterioration (TTD) by Quality of Life (QoL) | At 12,18 and 24 months
  CFB in the global health status (GHS) score and each scale of the EORTC QLQ-C30 questionnaire.
  Patient reported outcomes of health-related quality of life will be assessed using the EORTC QLQ-C30 questionnaire and analyzed on the QoL population.
  Published scoring manuals and guidelines will be used to generate scale scores and handle missing data. Descriptive statistics for actual values will be tabulated at each scheduled time point.
  TTD will be assessed using the Kaplan-Meier method. The median event time and 95% CI for the median will be estimated if reached. TTD will be censored at the date of the last QoL assessment prior to the start of a new therapy.
Incidence of Tolerability | Through study completion, an average of 58 months
  It will be assessed by incidence of different type of dose modifications, discontinuations due to AEs, number of administered cycles, etc.
Exposure levels of nadunolimab when administered in combination with gemcitabine plus carboplatin (Pharmacokinetics) | Days 1 and 8 from all cycles and post-treatment visit, an average of 58 months
  Blood samples for nadunolimab serum concentration analysis will be collected prior to each nadunolimab infusion and 1 hour after the end of each nadunolimab infusion on Day 1 and on Day 8 (all cycles), and at post-treatment visit (30 (±3) days after the last dose of study treatment.
Anti-drug antibodies (ADAs) against nadunolimab (Immunogenicity) | Days 1 and 8 from all cycles and post-treatment visit, an average of 58 months
  The formation of ADAs against nadunolimab will be assessed in blood samples collected prior to nadunolimab administration on Day 1 of each cycle and post-treatment visit.
  Immunogenicity will be evaluated by determination of the presence of ADAs as measured in serum by a tiered testing approach involving an initial screening assay, confirmation, and titration of confirmed positive samples. Samples will be banked so that further characterisation of the effect of ADAs upon nadunolimab binding to its target antigen may be undertaken.
  Characterisation of banked samples will include assessment of neutralising antibodies for samples that have been confirmed positive for ADA

CONTACTS AND LOCATIONS:
Overall Officials: Chief Investigator, Study Director — Hospital General Universitario Gregorio; Chief Investigator, Study Director — Clínica Universitaria de Navarra; Chief Investigator, Study Director — Instituto de Investigación Sanitaria (IIS) Biodonostia - OSI; Chief Medical Officer, Study Director — Cantargia AB
Locations (23):
- Spain (23):
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Universitario Clinico San Cecilio, Granada, Andalusia
  - Complejo Hospitalario de Jaén, Jaén, Andalusia
  - Hospital Universitario Virgen De La Victoria, Málaga, Andalusia
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitario Virgen Del Rocío, Seville, Andalusia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Onkologikoa, Donostia / San Sebastian, Basque Country
  - Complejo Hospitalario Universitario de Albacete, Albacete, Castille-La Mancha
  - Hospital Universitario de Toledo, Toledo, Castille-La Mancha
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - ICO Institut Catalá d'Oncologia de L´Hospitalet, Hospitalet de Llobregat, Barcelona, Catalonia
  - Hospital Universitario Arnau de Vilanova Lleida, Lleida, Catalonia
  - Complejo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Hospital Universitario Lucus Augusti, Lugo, Galicia
  - Hospital Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario San Juan de Alicante, Alicante, Valencia
  - Fundación Instituto Valenciano de Oncología, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol and the Statistical Analysis Plan (SAP) will be shared on the ClinicalTrials.gov web site. Also, results will be publish on congresses and manuscripts in scientific journal.
Supporting Information: Study Protocol
Time Frame: When results will be analyzed following the Statistical Analysis Plan (SAP).
Access Criteria: The results will be published. Every efforts Will be made to have open-access manuscripts.
URL: https://cantargia.com/

REFERENCES:
- See also: Description GEICAM is a Spanish Breast Cancer Research Group — http://www.geicam.org/